CLINICAL TRIAL: NCT04322604
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of AK002 in Patients With Moderately to Severely Active Eosinophilic Gastritis and/or Eosinophilic Duodenitis (Formerly Referred to as Eosinophilic Gastroenteritis)
Brief Title: A Study to Assess AK002 in Eosinophilic Gastritis and/or Eosinophilic Duodenitis (Formerly Referred to as Eosinophilic Gastroenteritis)
Acronym: ENIGMA 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK002-016
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Eosinophilic Gastritis; Eosinophilic Duodenitis
Keywords: Eosinophil; Eosinophilic; Eosinophilic gastrointestinal disorders; EGID; EG; EGE; Eosinophilic Gastritis; Eosinophilic Gastroenteritis; Eosinophilic Duodenitis
MeSH Terms: conditions — Eosinophilic enteropathy; Eosinophilic Esophagitis | interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 3 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive 6 monthly doses of lirentelimab (AK002): a first dose of 1 mg/kg followed by 5 monthly doses of 3 mg/kg.
  Interventions: Drug: lirentelimab (AK002)

INTERVENTIONS:
Drug: lirentelimab (AK002) — Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.
  Arms: 3 mg/kg of lirentelimab (AK002)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3, multi-center, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of lirentelimab (AK002), given monthly for 6 doses, in patients with moderately to severely active Eosinophilic Gastritis and/or Eosinophilic Duodenitis (formerly referred to as Eosinophilic Gastroenteritis) who have an inadequate response with, lost response to, or were intolerant to standard therapies

ELIGIBILITY:
Key Inclusion Criteria:

1. Provide written informed consent.
2. Male or female aged ≥18 and ≤80 years at the time of signing the informed consent for entry.
3. Baseline endoscopic biopsy with ≥30 eosinophils/hpf in 5 hpf in the stomach and/or ≥30 eosinophils/hpf in 3 hpf in the duodenum, as determined by central histology assessment of biopsies collected during the screening EGD.
4. Completion of at least 4 daily PRO questionnaires per week for a minimum of 3 weeks during screening.
5. Patients with inadequate or loss of response to, or who were intolerant to standard therapies for EG/EoD symptoms, which could include PPI, antihistamines, systemic or topical corticosteroids, and/or diet, among others.
6. If patient is on pre-existing dietary restrictions, willingness to maintain dietary restrictions throughout the study.
7. Willing and able to comply with all study procedures and visit schedule including follow-up visits.
8. Female patients must be either post-menopausal for at least 1 year with FSH level >30 mIU/mL at screening or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from screening until the end of the study, or for 120 days following the last dose of study drug, whichever is longer. Male patients with female partners of childbearing potential must agree to use a highly effective method of contraception from screening until the end of the study or for 120 days following the last dose of study drug, whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or later menstrual period) at any time during study participation.

Key Exclusion Criteria:

1. Use of systemic or topical corticosteroids exceeding the equivalent of 10 mg/day of prednisone within 4 weeks prior to the screening visit.
2. Change in the dose of corticosteroids (systemic or topical), PPI, leukotrienes, or diet therapy within 4 weeks prior to the screening visit.
3. Treatment with any immunosuppressive or immunomodulatory drugs that may interfere with the study within 12 weeks prior to the screening visit.
4. Prior exposure to AK002 or known hypersensitivity to any constituent of the study drug.
5. Active Helicobacter pylori infection, unless treated and confirmed to be negative prior to randomization and symptoms remain consistent.
6. History of inflammatory bowel disease, celiac disease, achalasia, or esophageal surgery.
7. History of bleeding disorders and/or esophageal varices.
8. Other causes of gastric and/or duodenal eosinophilia or eosinophilic granulomatosis with polyangiitis (EGPA).
9. Confirmed diagnosis of Hypereosinophilic Syndrome (HES).
10. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
11. Presence of an abnormal laboratory value considered to be clinically significant by the Investigator.
12. Any disease, condition (medical or surgical), or cardiac abnormality, which, in the opinion of the Investigator, would place the patient at increased risk.
13. History of malignancy, except carcinoma in situ, early stage prostate cancer, or non-melanoma skin cancers. However, cancers that have been in remission for more than 5 years and are considered cured, can be enrolled (with the exception of breast cancer).
14. Treatment for a clinically significant helminthic parasitic infection within 6 months of screening.
15. Positive Ova and Parasite (O&P) test and/or seropositive for Strongyloides stercoralis.
16. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected within 5 half-lives (4 months) of study drug administration.
17. Seropositive for HIV or hepatitis at screening, except for vaccinated patients or patients with past but resolved hepatitis, at screening.
18. Participation in a concurrent interventional study with the last intervention occurring within 30 days prior to study drug administration (or 90 days or 5 half-lives, whichever is longer, for biologic products).
19. Known history of alcohol, drug, or other substance abuse or dependence, considered by the Investigator to be ongoing and clinically significant.
20. Any other reason that in the opinion of the Investigator or the Medical Monitor makes the patient unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Paterson, MD, Study Director — Allakos Inc.
Locations (57):
- United States (57):
  - Allakos Investigational Site, Birmingham, Alabama
  - Allakos Investigational Site, Huntsville, Alabama
  - Allakos Investigational Site, Gilbert, Arizona
  - Allakos Investigational Site, Phoenix, Arizona
  - Allakos Investigational Site, Scottsdale, Arizona
  - Allakos Investigational Site, Little Rock, Arkansas
  - Allakos Investigational Site, Chula Vista, California
  - Allakos Investigational Site, La Jolla, California
  - Allakos Investigational Site, Murrieta, California
  - Allakos Investigational Site, Oakland, California
  - Allakos Investigational Site, Santa Monica, California
  - Allakos Investigational Site, Tustin, California
  - Allakos Investigational Site, Ventura, California
  - Allakos Investigational Site, Walnut Creek, California
  - Allakos Investigational Site, Aurora, Colorado
  - Allakos Investigational Site, Colorado Springs, Colorado
  - Allakos Investigational Site, Bristol, Connecticut
  - Allakos Investigational Site, Brandon, Florida
  - Allakos Investigational Site, Edgewater, Florida
  - Allakos Investigational Site, Jacksonville, Florida
  - Allakos Investigational Site, Miami, Florida
  - Allakos Investigational Site, New Port Richey, Florida
  - Allakos Investigational Site, Atlanta, Georgia
  - Allakos Investigational Site, Chicago, Illinois
  - Allakos Investigational Site, Crowley, Louisiana
  - Allakos Investigational Site, Chevy Chase, Maryland
  - Allakos Investigational Site, Boston, Massachusetts
  - Allakos Investigational Site, Ann Arbor, Michigan
  - Allakos Investigational Site, Rochester, Minnesota
  - Allakos Investigational Site, Kansas City, Missouri
  - Allakos Investigational Site, Las Vegas, Nevada
  - Allakos Investigational Site, Reno, Nevada
  - Allakos Investigational Site, Great Neck, New York
  - Allakos Investigational Site, New York, New York
  - Allakos Investigational Site, Chapel Hill, North Carolina
  - Allakos Investigational Site, Charlotte, North Carolina
  - Allakos Investigational Site, Durham, North Carolina
  - Allakos Investigational Site, Rocky Mount, North Carolina
  - Allakos Investigational Site, Cincinnati, Ohio
  - Allakos Investigational Site, Cleveland, Ohio
  - Allakos Investigational Site, Dayton, Ohio
  - Allakos Investigational Site, Mentor, Ohio
  - Allakos Investigational Site, Oklahoma City, Oklahoma
  - Allakos Investigational Site, Danville, Pennsylvania
  - Allakos Investigational Site, Philadelphia, Pennsylvania
  - Allakos Investigational Site, Chattanooga, Tennessee
  - Allakos Investigational Site, Hixson, Tennessee
  - Allakos Investigational Site, Kingsport, Tennessee
  - Allakos Investigational Site, Nashville, Tennessee
  - Allakos Investigational Site, Austin, Texas
  - Allakos Investigational Site, Houston, Texas
  - Allakos Investigational Site, Ogden, Utah
  - Allakos Investigational Site, Riverton, Utah
  - Allakos Investigational Site, Salt Lake City, Utah
  - Allakos Investigational Site, Sandy City, Utah
  - Allakos Investigational Site, Fairfax, Virginia
  - Allakos Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Started | 91 | 90
Completed | 85 | 83
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo | Total
Number analyzed (Participants) | 91 | 89 | 180
Age, Continuous [Median (Full Range); unit: years] | 43 [17 to 77] | 41 [18 to 78] | 42 [17 to 78]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 81 | 85 | 166
  >=65 years | 10 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 61 | 117
  Male | 35 | 28 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 24
  Not Hispanic or Latino | 76 | 78 | 154
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 7 | 6 | 13
  White | 75 | 78 | 153
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 89 | 180
Baseline Gastric Eosinophil Count [Mean (Standard Deviation); unit: Eosinophils/HPF] — Eosinophil Count (cells/HPF) in gastric tissue
  Eosinophils/HPF | 51.3 (57.9) | 37.0 (30.9) | 44.3 (46.9)
Baseline Duodenal Eosinophil Count [Mean (Standard Deviation); unit: Eosinophils/HPF] — Eosinophil Count (cells/HPF) in duodenal tissue Population: One subject did not have the duodenal biopsy samples
  Eosinophils/HPF
    number analyzed (Participants) | 91 | 88 | 179
    (all) | 42.4 (19.8) | 39.1 (15.6) | 40.7 (17.9)
Baseline Patient Reported Outcome Total and Symptom Scores [Mean (Standard Deviation); unit: Score on a scale] | 29.5 (11.0) | 27.7 (11.1) | 28.6 (11.0)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Tissue Eosinophil Responders at Week 24
Description: A tissue eosinophil responder is defined as mean eosinophil count ≤4 cells/HPF in 5 gastric HPFs for EG only patients, ≤15 cells/HPF in 3 duodenal HPFs for EoD only patients, and ≤4 cells/HPF in 5 gastric HPFs and ≤15 cells/HPF in 3 duodenal HPFs for EG+EoD patients.
Time Frame: At Week 24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 91 | 89
Participants | 77 | 4
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 80.1, 95% CI 2-sided [70.1 to 87.9]

2. Primary Outcome: Change in PRO Total Symptom Score (TSS) From Baseline to Weeks 23-24
Description: The PRO Total Symptom Score (TSS) is a patient reported outcome (PRO) questionnaire comprises the following 6 symptoms: Abdominal pain intensity, Nausea intensity, Fullness before meal intensity, Loss of appetite intensity, Bloating intensity, and Abdominal cramping intensity. TSS scores can range from 0 to 60, with a lower score indicating less-severe symptoms.
Time Frame: Baseline to Weeks 23 - 24
Population: Modified Intention-to-treat
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 91 | 89
Score on a scale | -10.0 (1.2) | -11.5 (1.1)
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.3427, ANCOVA; LSM Difference from Placebo = 1.5, 95% CI 2-sided [-1.6 to 4.7]

3. Secondary Outcome: Change in Tissue Eosinophils From Baseline to Week 24
Description: Tissue eosinophil count obtained in biopsy specimens from the stomach and/or duodenum using esophago-gastro-duodenoscopy (EGD)
Time Frame: Baseline to Week 24
Population: Modified Intention-to-treat
Measure: Mean (Standard Deviation); unit: Cells/HPF
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 83 | 83
Cells/HPF | -61.6 (46.3) | -11.7 (21.3)
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LSM Difference from Placebo = -41.2, 95% CI 2-sided [-48.1 to -34.2]

4. Secondary Outcome: Subjects Achieving Mean Eosinophil Count ≤1 Cell/Hpf in 5 Highest Gastric Hpf and/or Mean Eosinophil Count ≤1 Cell/Hpf in 3 Highest Duodenal Hpf at Week 24
Description: as for outcome 3
Time Frame: At Week 24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 91 | 89
Participants | 75 | 1
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 81.3, 95% CI 2-sided [71.7 to 88.8]

5. Secondary Outcome: Number of Treatment Responders
Description: Treatment responders defined by >30% improvement in TSS at Weeks 23-24 and eosinophil count ≤4 cells/hpf in 5 gastric hpf and/or eosinophil count ≤15 cells/hpf in 3 duodenal hpf at Week 24
Time Frame: Weeks 23-24 and at Week 24, respectively
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 91 | 89
Participants | 39 | 3
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 39.5, 95% CI 2-sided [25.4 to 52.2]

6. Secondary Outcome: Subjects Who Achieve ≥50% Reduction in TSS From Baseline to Weeks 23-24
Description: as for outcome 2
Time Frame: At Weeks 23-24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 91 | 89
Participants | 36 | 29
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.3549, Fisher Exact; Percent Difference from Placebo = 7.0, 95% CI 2-sided [-7.4 to 21.6]

7. Secondary Outcome: Subjects Who Achieve ≥70% Reduction in TSS From Baseline to Weeks 23-24
Description: as for outcome 2
Time Frame: At Weeks 23-24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 91 | 89
Participants | 26 | 18
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.2262, Fisher Exact; Percent Difference from Placebo = 8.3, 95% CI 2-sided [-6.3 to 22.7]

8. Secondary Outcome: Percent Change in Weekly TSS Over Time Using MMRM
Description: as for outcome 2
Time Frame: Baseline to Week 24
Population: Modified Intention-to-treat
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 91 | 89
Percentage of Change
  Week 2 | -18.2 (34.1) | -17.4 (31.9)
  Week 4 | -17.7 (34.2) | -21.2 (32.8)
  Week 6 | -29.8 (37.2) | -28.3 (37.6)
  Week 8 | -29.8 (40.4) | -31.3 (33.6)
  Week 10 | -34.6 (39.7) | -36.3 (39.7)
  Week 12 | -33.1 (39.9) | -36.2 (37.3)
  Week 14 | -36.3 (40.2) | -38.7 (36.5)
  Week 16 | -33.1 (40.8) | -38.8 (38.8)
  Week 18 | -42.6 (42.3) | -41.3 (37.2)
  Week 20 | -42.1 (37.1) | -39.9 (34.9)
  Week 22 | -41.7 (39.8) | -41.4 (37.3)
  Week 24 | -39.4 (39.9) | -38.5 (37.2)
Statistical Analysis 1: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Week 24 Percent Change from Baseline; Test type: Superiority; p = 0.3812, Mixed Models Analysis; LSM Difference from Placebo = 5.0, 95% CI 2-sided [-6.1 to 16.0]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 225
Arm/Group | 3 mg/kg of Lirentelimab (AK002) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/89
Serious Adverse Events (participants affected / at risk) | 7/91 | 5/89
Other Adverse Events (participants affected / at risk) | 41/91 | 31/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg/kg of Lirentelimab (AK002) (N=91) | Placebo (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg/kg of Lirentelimab (AK002) (N=91) | Placebo (N=89)
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 5 | 1
Corona virus infection (Infections and infestations) | 4 | 6
Urinary tract infection (Infections and infestations) | 3 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 31 | 12
Coronavirus test positive (Investigations) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (2):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT04322604/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT04322604/SAP_001.pdf